CLINICAL TRIAL: NCT04545814
Title: A Pilot Study Analyzing Preoperative Stereotactic Radiosurgery (SRS) With Gamma Knife (GK) for Brain Metastases
Brief Title: Analyzing Preoperative Stereotactic Radiosurgery With Gamma Knife Icon for Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Straza, MD, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038835
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
Keywords: brain metastases; Gamma Knife; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental): SRS will be delivered utilizing gamma knife or linear accelerator-based techniques.
  Interventions: Device: Stereotactic Radiosurgery

INTERVENTIONS:
Device: Stereotactic Radiosurgery — Maximum Tumor Diameter ≤ 2 cm = 20-24 Gy; Maximum Tumor Diameter 2.1-3.0 cm = 18 Gy; Maximum Tumor Diameter 3.1-5.0 cm = 15 Gy
  Other Names: SRS

SUMMARY:
This is a single-arm, single-center pilot study in which 10 patients with one to four brain metastases diagnosed on brain magnetic resonance imaging (MRI) within the past 30 days will be evaluated for study eligibility and enrolled as appropriate.

DETAILED DESCRIPTION:
INTERVENTION: Enrolled patients will receive stereotactic radiosurgery (SRS) to all metastases followed by surgical resection of resectable metastases within one to 10 days following SRS. Pathologic specimens will be analyzed, and the patient will enter a standard pattern of surveillance (brain MRI every three months for two years).

STUDY RATIONALE: Given the increased risk of leptomeningeal failure with surgery followed by SRS as well as the risk of radiation necrosis, new paradigms in therapy delivery and sequencing are being explored. Areas of investigation include optimization of target volume, marginal expansion, multi-fractionation, timeliness of SRS after surgery, and delivery of SRS prior to surgical resection. In theory, advantages of preoperative SRS include better target delineation, sterilization of tumor cells prior to surgical disruption of the tumor, vascular supply, and CSF spaces, and resection of tissue that would otherwise be at risk of radiation necrosis.

In 2014, Asher, et al. (Asher AL, Burri SH, Wiggins WF, et al. A new treatment paradigm: neoadjuvant radiosurgery before surgical resection of brain metastases with analysis of local tumor recurrence. Int J Radiat Oncol Biol Phys 2014;88:899-906.) reported that the use of neoadjuvant SRS prior to surgery was both safe and effective (even for metastases >3 cm) with no reported leptomeningeal recurrences or radiation necrosis. More recently, Patel et al. (Patel KR, Burri SH, Asher AL, et al. Comparing Preoperative With Postoperative Stereotactic Radiosurgery for Resectable Brain Metastases: A Multi-institutional Analysis. Neurosurgery 2016;79:279-85.) performed a retrospective comparison of preoperative versus postoperative SRS and reported no difference in local control, distant brain failure, or overall survival. Furthermore, the authors reported significantly lower rates of leptomeningeal carcinomatosis and radiation necrosis with preoperative SRS.

Huff, et al. (Huff WX, Agrawal N, Shapiro S, et al. Efficacy of pre-operative stereotactic radiosurgery followed by surgical resection and correlative radiobiological analysis for patients with 1-4 brain metastases: study protocol for a phase II trial. Radiat Oncol 2018;13:252.) recently published a protocol for a phase II prospective trial designed to compare outcomes using preoperative SRS versus historically cited outcomes for postoperative SRS. This pilot study mirrors this design and aims to confirm study feasibility and to assess local control, central nervous system (CNS) progression-free survival, overall survival, rates of leptomeningeal spread, rates of radiation necrosis, and quality of life measures with the use of preoperative SRS.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study related procedure that's is not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Female or Male subject's ≥ 18 years old at the time of informed consent.
3. Radiographically confirmed solid tumor brain metastases.
4. Criteria for surgical resection of at least one metastasis per neurosurgeon discretion.
5. Stereotactic radiosurgery candidate per radiation oncologist discretion.
6. A diagnostic MRI Brain or CT Head demonstrating the presence of 1-4 solid tumor brain metastases and lesion to be resected no more than 5 cm in any direction, performed within 30 days prior to stereotactic radiosurgery.
7. For known and unknown primary, diagnosis-specific graded prognostic assessment (ds-GPA) estimated median survival no less than 6 months.
8. Surgical resection able to be performed within 1-10 days after radiosurgery.
9. Patients currently on cytotoxic chemotherapy or immunotherapy are eligible, not including anti-vascular endothelial growth factor (anti-VEGF) therapy.
10. Female subjects who:

    1. Are postmenopausal for at least 1 year before the screening visit, OR
    2. Are surgically sterile, OR

    i. Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last study Intervention (female and male condoms should not be used together), OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
11. Male subjects, even if surgically sterilized (ie, status post-vasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through 4 months after the last study Intervention (female and male condoms should not be used together), OR
    2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

1. Patients who received anti-VEGF therapy within 6 weeks prior to enrollment, as there is increased risk of fatal brain hemorrhage with surgical resection.
2. Major medical illnesses or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and/or interfere with surveillance.
3. Patients with more than 4 brain metastases on MRI Brain.
4. Lesion to be resected is more than 5 cm in any dimension.
5. Patients with leptomeningeal metastases documented by MRI or cerebrospinal fluid (CSF) evaluation.
6. Previous whole brain radiation therapy.
7. Previous radiation therapy to the lesion to be resected.
8. Planned adjuvant focal therapy including additional radiation therapy to the brain.
9. Not a surgical candidate per neurosurgeon discretion.
10. Not a stereotactic radiosurgery candidate per radiation oncologist discretion.
11. Surgery unable to be performed between 1 - 10 days after radiosurgery.
12. Women who are pregnant or nursing as treatment involves unforeseeable risks to the fetus or child.
13. Patients who have a known or unknown primary and have an estimated median survival of less than 6 months per ds-GPA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
The number of subjects undergoing resection following SRS. | 10 days following SRS
  All subjects undergoing resection following SRS will be documented.
The number of subjects with no identifiable disease following resection. | 20 months
  Identifiable disease will be determined by post-treatment MRI of the brain.

SECONDARY OUTCOMES:
The number of subjects achieving CNS progression-free survival. | 6, 12 and 18 months
  This will be measured using the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. Subjects will be evaluated at six, 12 and 18 months.
The number of subjects achieving overall survival. | 6, 12 and 18 months
  The number of subjects alive at six, 12 and 18 months following surgical resection.
The number of subjects with leptomeningeal carcinomatosis using preoperative SRS. | Two years
  The number of subjects with this diagnosis will be documented.
The number of subjects with radiation necrosis. | Two years
  Radiation necrosis will be determined by radiographic appearance on posttreatment MRI. The number of patients with radiation necrosis will be documented.
The number of subjects reporting a high quality of life. | Every 3 months until two years
  Quality of life will be measured by the MD Anderson Symptom Inventory for brain tumor (MDASI-BT). The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 numeric rating scale (NRS), with 0 being "not present" and 10 being "as bad as you can imagine."

CONTACTS AND LOCATIONS:
Overall Officials: Michael Straza, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asher AL, Burri SH, Wiggins WF, Kelly RP, Boltes MO, Mehrlich M, Norton HJ, Fraser RW. A new treatment paradigm: neoadjuvant radiosurgery before surgical resection of brain metastases with analysis of local tumor recurrence. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):899-906. doi: 10.1016/j.ijrobp.2013.12.013. PMID 24606851
- [Background] Patel KR, Burri SH, Asher AL, Crocker IR, Fraser RW, Zhang C, Chen Z, Kandula S, Zhong J, Press RH, Olson JJ, Oyesiku NM, Wait SD, Curran WJ, Shu HK, Prabhu RS. Comparing Preoperative With Postoperative Stereotactic Radiosurgery for Resectable Brain Metastases: A Multi-institutional Analysis. Neurosurgery. 2016 Aug;79(2):279-85. doi: 10.1227/NEU.0000000000001096. PMID 26528673
- [Background] Huff WX, Agrawal N, Shapiro S, Miller J, Kulwin C, Shah M, Savage JJ, Payner T, Vortmeyer A, Watson G, Dey M. Efficacy of pre-operative stereotactic radiosurgery followed by surgical resection and correlative radiobiological analysis for patients with 1-4 brain metastases: study protocol for a phase II trial. Radiat Oncol. 2018 Dec 20;13(1):252. doi: 10.1186/s13014-018-1178-8. PMID 30572923

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04545814/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04545814/ICF_001.pdf